CLINICAL TRIAL: NCT06183853
Title: Evaluation of the Long-term Results of Extended Supra-basillary Genioplasty of the "Chin Wing" Type Without Bone Graft: Aesthetic and Functional Satisfaction, Sensory Recovery and Bone Healing
Brief Title: Evaluation of the Long-term Results of Extended Supra-basillary Genioplasty of the "Chin Wing" Type Without Bone Graft
Acronym: SASCWatch
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8702
Record Dates: First submitted 2022-09-14; First posted 2023-12-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-12

CONDITIONS: Maxillofacial Abnormalities
Keywords: Dysmorphoses; Maxillofacial Abnormalities; Maxillomandibular; Lip incompetence; Ventilation disorders; Genioplasty
MeSH Terms: conditions — Maxillofacial Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The correction of maxillomandibular dysmorphoses, responsible for both functional discomfort (lip incompetence, ventilation disorders, periodontal disease) but also aesthetic, calls in particular for genioplasty, of which there are several techniques. One of these chin repositioning techniques, called "Chin Wing", cuts the bone to optimize the functional and aesthetic result. While all genioplasty techniques expose the risk of nerve damage and lack of bone consolidation, these parameters are only rarely addressed in the literature in the specific context of this extensive bone cutting.

The objective of this work is to assess the satisfaction of patients who have benefited from chin advancement surgery using the "Chin Wing" technique.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 18 years old)
* having undergone "Chin Wing" type genioplasty surgery in the maxillofacial surgery department of Strasbourg between October 1, 2012 and June 30, 2022.
* Subject who has not expressed his opposition to the reuse of his data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed their opposition to the reuse of their data for scientific research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) having undergone "Chin Wing" type genioplasty surgery in the maxillofacial surgery department of Strasbourg between October 1, 2012 and June 30, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Aesthetic and functional satisfaction of the patients' results of surgery | 6 months after surgery
  Aesthetic and functional satisfaction of the patients who have benefited from chin advancement surgery using the "Chin Wing" technique.
  This satisfaction is assessed by a satisfaction questionnaire of 10 questions. Single answer out of 4 items proposed per question.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Plastique, Reconstructrice, Esthétique et Maxillo-faciale - CHU de Strasbourg - France, Strasbourg, France